CLINICAL TRIAL: NCT00004562
Title: Occluded Artery Trial (OAT) - Randomized Comparative Effectiveness Trial of PCI and Medical Therapy Only Post MI
Brief Title: Occluded Artery Trial (OAT)
Acronym: OAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130; U01HL062509-01A1 (NIH)
Record Dates: First submitted 2000-02-09; First posted 2000-02-10 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Heart Failure | interventions — Adrenergic beta-Antagonists; Platelet Aggregation Inhibitors; Stents; Angioplasty, Balloon, Coronary; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal Medical Therapy Only (MED) (Active Comparator): Conventional medical management, including aspirin, beta blockers, angiotensin converting enzyme (ACE) inhibitors, and risk factor modification
  Interventions: Drug: Beta adrenergic blockers; Drug: Platelet inhibitors; Drug: ACE Inhibitors
- Percutaneous Coronary Intervention (PCI) (Experimental): Conventional medical management, including aspirin, beta blockers, angiotensin converting enzyme (ACE) inhibitors, and risk factor modification, plus percutaneous coronary intervention and coronary stenting
  Interventions: Drug: Beta adrenergic blockers; Drug: Platelet inhibitors; Procedure: PTCA and stents; Drug: ACE Inhibitors

INTERVENTIONS:
Drug: Beta adrenergic blockers — Participants will receive beta adrenergic blockers.
  Other Names: beta blockers
Drug: Platelet inhibitors — Participants will receive platelet inhibitors.
  Other Names: Antiplatelet drugs
Procedure: PTCA and stents — Participants will undergo percutaneous coronary intervention (PTCA) and coronary stenting.
  Other Names: Percutaneous Transluminal Coronary Angioplasty; and; Stent Placement
  Arms: Percutaneous Coronary Intervention (PCI)
Drug: ACE Inhibitors — Participants will receive ACE inhibitors.
  Other Names: angiotensin-converting-enzyme inhibitor

SUMMARY:
The purpose of this study is to determine whether opening an occluded infarcted artery 3-28 days after an acute myocardial infarction in high-risk asymptomatic patients reduces the composite endpoint of mortality, recurrent myocardial infarction, and hospitalization for class IV congestive heart failure over an average 2.9-year follow-up with extended follow up for an average of six years. Long term follow-up of patients were completed in March 2010. Final collection of all regulatory documentation was completed June 2011.

DETAILED DESCRIPTION:
BACKGROUND:

The benefits of establishing early coronary reperfusion in acute myocardial infarction (MI) have now been unequivocally established. However, current pharmacologic strategies fail to achieve effective reperfusion in 30 percent or more of patients, and many patients with occluded infarct arteries do not meet current criteria for use of these agents. Early angioplasty, an effective reperfusion method, is available to a small proportion of potentially eligible US acute MI patients. Hence a substantial number of acute MI patients pass the time when reperfusion therapy has any documented benefit (12 - 24 hours) with a persistently closed infarct vessel. Several lines of experimental and clinical evidence suggest that late reperfusion of these patients could provide clinically significant reductions in mortality and morbidity.

DESIGN NARRATIVE:

Multicenter, randomized, controlled. Patients at 217 clinical sites in the United States, Canada and Internationally were randomly allocated to two treatment arms over five years. One treatment consists of conventional medical management including aspirin, beta blockers, angiotensin converting enzyme (ACE) inhibitors, and risk factor modification. The other treatment consists of conventional medical therapy plus percutaneous coronary intervention and coronary stenting. Clinical outcomes will be compared using an intention-to-treat analysis. The primary composite endpoint is mortality, recurrent myocardial infarction, and hospitalization for NYHA Class IV congestive heart failure over a three year follow-up. Individual components of the study composite primary endpoint will be compared in the two treatment arms, as will the medical costs of the two treatments and the health-related quality of life. The cost-effectiveness of percutaneous revascularization will be assessed in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Recent MI (3-28 days) (Day 1 is the calendar day of the MI system onset)
* MI is defined based on at least 2 of 3 MI criteria confirmed by: 1) ischemic symptoms ≥30 minutes, 2) cardiac serum marker elevation (creatine kinase (CK) ≥2x upper limit of normal and CK-MB elevated above the upper limit of the laboratory normal) or troponin T, or troponin I elevated at least twice the upper limit of normal, 3) EKG: New Q-waves of ≥0.03 sec and/or 1/3 of QRS complex in ≥2 related EKG leads. If cardiac serum markers are elevated (2), any one of the following EKG findings satisfy inclusion criteria; new ST-T changes (ST elevation or depression), new left bundle-branch block (LBBB), loss of R-wave voltage ≥50% in ≥2 related leads or deep T wave inversions ≥3mm in ≥2 leads.
* TIMI flow 0 or 1 in infarct related artery (IRA)
* Meets criteria for high risk: EF <50% or site of occlusion is proximal, in left anterior descending (proximal to the second major diagonal branch); large right coronary artery; or circumflex, if supplying large obtuse marginal, and part of inferior wall (i.e., large dominant or co-dominant vessel).

Exclusion Criteria:

* Age <18 y
* Clinical indication for revascularization defined as follows: rest or low-threshold angina after MI; severe inducible ischemia on low level exercise or pharmacological stress testing (ST decreased ≥2 mm or inability to complete stage 1 or achieve 3-4 metabolic equivalents without angina, hypotension, or reversible perfusion defects in multiple territories or decreased wall motion thickening in >2 segments on echocardiogram); left main coronary disease (≥50% stenosis); or triple-vessel disease (3 major epicardial coronaries with >70% stenoses)
* Serious illness such as cancer or pulmonary disease that limits 3-year survival
* Severe renal disease defined as serum creatinine >3.0 mg/dL that markedly increases risk of radiographic contrast
* Severe valvular disease
* History of anaphylaxis to radiographic contrast
* Infarct artery too small (reference segment diameter <2.5 mm), target segment within or beyond extreme tortuosity (>90° angulation), or otherwise technically a poor candidate for PCI
* Chronic occlusion of IRA (seen on angiogram obtained before index MI or angiographic evidence of chronicity, e.g., presence of bridging collaterals)
* NYHA classes III-IV CHF; patients may be treated for acute heart failure complicating MI and rescreened
* Cardiogenic shock or sustained hypotension: systolic BP <90 mm Hg or cardiac index <2.2 L/min per m^2
* LV aneurysm in the same location as index MI and present before index MI
* Inability to cooperate with the protocol
* Patient refusal or inability to give informed consent
* Refusal of patient's physician to allow patient to participate
* Pregnancy
* Contraindication to anticoagulation during PCI or to routine antiplatelet therapy after stent implantation
* Qualifying IRA that has been grafted previously; patients with prior CABG may be enrolled if the IRA was not previously grafted
* Dilated or hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2201 (Actual)
Dates: Start 1999-09; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Hochman, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Hochman JS, Lamas GA, Knatterud GL, Buller CE, Dzavik V, Mark DB, Reynolds HR, White HD; Occluded Artery Trial Research Group. Design and methodology of the Occluded Artery Trial (OAT). Am Heart J. 2005 Oct;150(4):627-42. doi: 10.1016/j.ahj.2005.07.002. PMID 16209957
- [Background] Skolnick AH, Reynolds HR, White HD, Menon V, Carvalho AC, Maggioni AP, Pearte CA, Gruberg L, Azevedo RE, Schroeder E, Forman SA, Lamas GA, Hochman JS, Dzavik V. Comparison of late results of percutaneous coronary intervention among stable patients </=65 versus >65 years of age with an occluded infarct related artery (from the Occluded Artery Trial). Am J Cardiol. 2012 Mar 1;109(5):614-9. doi: 10.1016/j.amjcard.2011.10.015. Epub 2011 Dec 14. PMID 22172242
- [Background] Deyell MW, Buller CE, Miller LH, Wang TY, Dai D, Lamas GA, Srinivas VS, Hochman JS. Impact of National Clinical Guideline recommendations for revascularization of persistently occluded infarct-related arteries on clinical practice in the United States. Arch Intern Med. 2011 Oct 10;171(18):1636-43. doi: 10.1001/archinternmed.2011.315. Epub 2011 Jul 11. PMID 21747002
- [Background] Udelson JE, Pearte CA, Kimmelstiel CD, Kruk M, Kufera JA, Forman SA, Teresinska A, Bychowiec B, Marin-Neto JA, Hochtl T, Cohen EA, Caramori P, Busz-Papiez B, Adlbrecht C, Sadowski ZP, Ruzyllo W, Kinan DJ, Lamas GA, Hochman JS. The Occluded Artery Trial (OAT) Viability Ancillary Study (OAT-NUC): influence of infarct zone viability on left ventricular remodeling after percutaneous coronary intervention versus optimal medical therapy alone. Am Heart J. 2011 Mar;161(3):611-21. doi: 10.1016/j.ahj.2010.11.020. PMID 21392619
- [Background] Devlin G, Reynolds HR, Mark DB, Rankin JM, Carvalho AC, Vozzi C, Sopko G, Caramori P, Dzavik V, Ragosta M, Forman SA, Lamas GA, Hochman JS. Loss of short-term symptomatic benefit in patients with an occluded infarct artery is unrelated to non-protocol revascularization: results from the Occluded Artery Trial (OAT). Am Heart J. 2011 Jan;161(1):84-90. doi: 10.1016/j.ahj.2010.09.009. PMID 21167338
- [Background] Steigen TK, Buller CE, Mancini GB, Jorapur V, Cantor WJ, Rankin JM, Thomas B, Webb JG, Kronsberg SS, Atchison DJ, Lamas GA, Hochman JS, Dzavik V. Myocardial perfusion grade after late infarct artery recanalization is associated with global and regional left ventricular function at one year: analysis from the Total Occlusion Study of Canada-2. Circ Cardiovasc Interv. 2010 Dec;3(6):549-55. doi: 10.1161/CIRCINTERVENTIONS.109.918722. Epub 2010 Nov 9. PMID 21062997
- [Background] Jorapur V, Lamas GA, Sadowski ZP, Reynolds HR, Carvalho AC, Buller CE, Rankin JM, Renkin J, Steg PG, White HD, Vozzi C, Balcells E, Ragosta M, Martin CE, Srinivas VS, Wharton Iii WW, Abramsky S, Mon AC, Kronsberg SS, Hochman JS. Renal impairment and heart failure with preserved ejection fraction early post-myocardial infarction. World J Cardiol. 2010 Jan 26;2(1):13-8. doi: 10.4330/wjc.v2.i1.13. PMID 20885993
- [Background] Steg PG, Kerner A, Mancini GB, Reynolds HR, Carvalho AC, Fridrich V, White HD, Forman SA, Lamas GA, Hochman JS, Buller CE; OAT Investigators. Impact of collateral flow to the occluded infarct-related artery on clinical outcomes in patients with recent myocardial infarction: a report from the randomized occluded artery trial. Circulation. 2010 Jun 29;121(25):2724-30. doi: 10.1161/CIRCULATIONAHA.109.933200. Epub 2010 Jun 14. PMID 20547926
- [Background] Kruk M, Buller CE, Tcheng JE, Dzavik V, Menon V, Mancini GB, Forman SA, Kurray P, Busz-Papiez B, Lamas GA, Hochman JS. Impact of left ventricular ejection fraction on clinical outcomes over five years after infarct-related coronary artery recanalization (from the Occluded Artery Trial [OAT]). Am J Cardiol. 2010 Jan 1;105(1):10-6. doi: 10.1016/j.amjcard.2009.08.644. PMID 20102883
- [Background] Buller CE, Rankin JM, Carere RG, Buszman PE, Pfisterer ME, Dzavik V, Thomas B, Forman S, Ruzyllo W, Mancini GB, Michalis LK, Abreu PF, Lamas GA, Hochman JS. Percutaneous coronary intervention in the Occluded Artery Trial: procedural success, hazard, and outcomes over 5 years. Am Heart J. 2009 Sep;158(3):408-15. doi: 10.1016/j.ahj.2009.05.035. PMID 19699864
- [Background] Malek LA, Reynolds HR, Forman SA, Vozzi C, Mancini GB, French JK, Dziarmaga M, Renkin JP, Kochman J, Lamas GA, Hochman JS. Late coronary intervention for totally occluded left anterior descending coronary arteries in stable patients after myocardial infarction: Results from the Occluded Artery Trial (OAT). Am Heart J. 2009 Apr;157(4):724-32. doi: 10.1016/j.ahj.2008.12.008. PMID 19332202
- [Background] Dzavik V, Buller CE, Devlin G, Carere RG, Mancini GB, Cantor WJ, Buszman PE, Rankin JM, Vozzi C, Ross JR, Forman S, Barton BA, Lamas AG, Hochman JS. Angiographic and clinical outcomes of drug-eluting versus bare metal stent deployment in the Occluded Artery Trial. Catheter Cardiovasc Interv. 2009 May 1;73(6):771-9. doi: 10.1002/ccd.21930. PMID 19309733
- [Background] Mark DB, Pan W, Clapp-Channing NE, Anstrom KJ, Ross JR, Fox RS, Devlin GP, Martin CE, Adlbrecht C, Cowper PA, Ray LD, Cohen EA, Lamas GA, Hochman JS; Occluded Artery Trial Investigators. Quality of life after late invasive therapy for occluded arteries. N Engl J Med. 2009 Feb 19;360(8):774-83. doi: 10.1056/NEJMoa0805151. PMID 19228620
- [Background] Kruk M, Kadziela J, Reynolds HR, Forman SA, Sadowski Z, Barton BA, Mark DB, Maggioni AP, Leor J, Webb JG, Kapeliovich M, Marin-Neto JA, White HD, Lamas GA, Hochman JS. Predictors of outcome and the lack of effect of percutaneous coronary intervention across the risk strata in patients with persistent total occlusion after myocardial infarction: Results from the OAT (Occluded Artery Trial) study. JACC Cardiovasc Interv. 2008 Oct;1(5):511-20. doi: 10.1016/j.jcin.2008.08.007. PMID 19194534
- [Background] Rashba EJ, Lamas GA, Couderc JP, Hollist SM, Dzavik V, Ruzyllo W, Fridrich V, Buller CE, Forman SA, Kufera JA, Carvalho AC, Hochman JS; OAT-EP Investigators. Electrophysiological effects of late percutaneous coronary intervention for infarct-related coronary artery occlusion: the Occluded Artery Trial-Electrophysiological Mechanisms (OAT-EP). Circulation. 2009 Feb 17;119(6):779-87. doi: 10.1161/CIRCULATIONAHA.108.808626. Epub 2009 Feb 2. PMID 19188505
- [Background] Menon V, Pearte CA, Buller CE, Steg PG, Forman SA, White HD, Marino PN, Katritsis DG, Caramori P, Lasevitch R, Loboz-Grudzien K, Zurakowski A, Lamas GA, Hochman JS. Lack of benefit from percutaneous intervention of persistently occluded infarct arteries after the acute phase of myocardial infarction is time independent: insights from Occluded Artery Trial. Eur Heart J. 2009 Jan;30(2):183-91. doi: 10.1093/eurheartj/ehn486. Epub 2008 Nov 21. PMID 19028780
- [Background] Jorapur V, Steigen TK, Buller CE, Dzavik V, Webb JG, Strauss BH, Yeoh EE, Kurray P, Sokalski L, Machado MC, Kronsberg SS, Lamas GA, Hochman JS, Mancini GB. Distribution and determinants of myocardial perfusion grade following late mechanical recanalization of occluded infarct-related arteries postmyocardial infarction: a report from the occluded artery trial. Catheter Cardiovasc Interv. 2008 Nov 15;72(6):783-9. doi: 10.1002/ccd.21745. PMID 18798327
- [Background] Lamas GA, Hochman JS. Where does the Occluded Artery Trial leave the late open artery hypothesis? Heart. 2007 Nov;93(11):1319-21. doi: 10.1136/hrt.2007.123489. PMID 17933981
- [Background] Lang IM, Forman SA, Maggioni AP, Ruzyllo W, Renkin J, Vozzi C, Steg PG, Hernandez-Garcia JM, Zmudka K, Jimenez-Navarro M, Sopko G, Lamas GA, Hochman JS. Causes of death in early MI survivors with persistent infarct artery occlusion: results from the Occluded Artery Trial (OAT). EuroIntervention. 2009 Nov;5(5):610-8. doi: 10.4244/eijv5i5a98. PMID 20142183
- [Background] Cantor WJ, Baptista SB, Srinivas VS, Pearte CA, Menon V, Sadowski Z, Ross JR, Meciar P, Nikolsky E, Forman SA, Lamas GA, Hochman JS. Impact of stress testing before percutaneous coronary intervention or medical management on outcomes of patients with persistent total occlusion after myocardial infarction: analysis from the occluded artery trial. Am Heart J. 2009 Apr;157(4):666-72. doi: 10.1016/j.ahj.2008.12.004. Epub 2009 Feb 23. PMID 19332193
- [Background] Sadanandan S, Buller C, Menon V, Dzavik V, Terrin M, Thompson B, Lamas G, Hochman JS. The late open artery hypothesis--a decade later. Am Heart J. 2001 Sep;142(3):411-21. doi: 10.1067/mhj.2001.117774. PMID 11526353
- [Background] Reynolds HR, Forman SA, Tamis-Holland JE, Steg PG, Mark DB, Pearte CA, Carvalho AC, Sopko G, Liu L, Lamas GA, Kruk M, Loboz-Grudzien K, Ruzyllo W, Hochman JS. Relationship of female sex to outcomes after myocardial infarction with persistent total occlusion of the infarct artery: analysis of the Occluded Artery Trial (OAT). Am Heart J. 2012 Mar;163(3):462-9. doi: 10.1016/j.ahj.2012.01.005. PMID 22424018
- [Background] White HD, Reynolds HR, Carvalho AC, Pearte CA, Liu L, Martin CE, Knatterud GL, Dzavik V, Kruk M, Steg PG, Cantor WJ, Menon V, Lamas GA, Hochman JS. Reinfarction after percutaneous coronary intervention or medical management using the universal definition in patients with total occlusion after myocardial infarction: results from long-term follow-up of the Occluded Artery Trial (OAT) cohort. Am Heart J. 2012 Apr;163(4):563-71. doi: 10.1016/j.ahj.2012.01.016. PMID 22520521
- [Background] Freixa X, Dzavik V, Forman SA, Rankin JM, Buller CE, Cantor WJ, Ruzyllo W, Reynolds HR, Lamas GA, Hochman JS. Long-term outcomes after a strategy of percutaneous coronary intervention of the infarct-related artery with drug-eluting stents or bare metal stents vs medical therapy alone in the Occluded Artery Trial (OAT). Am Heart J. 2012 Jun;163(6):1011-8. doi: 10.1016/j.ahj.2012.03.008. PMID 22709754
- [Background] Hastings RS, Hochman JS, Dzavik V, Lamas GA, Forman SA, Schiele F, Michalis LK, Nikas D, Jaroch J, Reynolds HR. Effect of late revascularization of a totally occluded coronary artery after myocardial infarction on mortality rates in patients with renal impairment. Am J Cardiol. 2012 Oct 1;110(7):954-60. doi: 10.1016/j.amjcard.2012.05.024. Epub 2012 Jun 22. PMID 22728005
- [Result] Hochman JS, Lamas GA, Buller CE, Dzavik V, Reynolds HR, Abramsky SJ, Forman S, Ruzyllo W, Maggioni AP, White H, Sadowski Z, Carvalho AC, Rankin JM, Renkin JP, Steg PG, Mascette AM, Sopko G, Pfisterer ME, Leor J, Fridrich V, Mark DB, Knatterud GL; Occluded Artery Trial Investigators. Coronary intervention for persistent occlusion after myocardial infarction. N Engl J Med. 2006 Dec 7;355(23):2395-407. doi: 10.1056/NEJMoa066139. Epub 2006 Nov 14. PMID 17105759
- [Result] Hochman JS, Reynolds HR, Dzavik V, Buller CE, Ruzyllo W, Sadowski ZP, Maggioni AP, Carvalho AC, Rankin JM, White HD, Goldberg S, Forman SA, Mark DB, Lamas GA; Occluded Artery Trial Investigators. Long-term effects of percutaneous coronary intervention of the totally occluded infarct-related artery in the subacute phase after myocardial infarction. Circulation. 2011 Nov 22;124(21):2320-8. doi: 10.1161/CIRCULATIONAHA.111.041749. Epub 2011 Oct 24. PMID 22025606
- [Derived] Xing Z, Pei J, Huang J, Hu X, Gao S. Relationship of obesity to adverse events in myocardial infarction patients without primary percutaneous coronary intervention: results from the Occluded Artery Trial (OAT). Curr Med Res Opin. 2019 Sep;35(9):1563-1569. doi: 10.1080/03007995.2019.1603993. Epub 2019 May 10. PMID 30950656
- [Derived] Jhaveri RR, Reynolds HR, Katz SD, Jeger R, Zinka E, Forman SA, Lamas GA, Hochman JS. Heart failure in post-MI patients with persistent IRA occlusion: prevalence, risk factors, and the long-term effect of PCI in the Occluded Artery Trial (OAT). J Card Fail. 2012 Nov;18(11):813-21. doi: 10.1016/j.cardfail.2012.10.012. PMID 23141853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The primary analysis of the trial included 2166 patients who had been enrolled through December 2005 with an average follow-up of 2.9 years. An additional 35 patients were enrolled through June 2006 during an extended period of enrollment in the nuclear viability ancillary study. All 2201 patients are included here.
Groups:
- Percutaneous Coronary Intervention Group: Percutaneous Coronary Intervention with stent placement and optimal medical therapy
- Medical Therapy Group: Conventional medical management, including aspirin, beta blockers, angiotensin converting enzyme (ACE) inhibitors, and risk factor modification, plus percutaneous coronary intervention and coronary stenting
Period: Overall Study
Arm/Group | Percutaneous Coronary Intervention Group | Medical Therapy Group
Started | 1101 | 1100
Completed | 999 | 1009
Not Completed | 102 | 91
Not completed — Lost to Follow-up | 102 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Coronary Intervention Group | Medical Therapy Group | Total
Number analyzed (Participants) | 1101 | 1100 | 2201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (10.9) | 58.7 (11.1) | 58.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 242 | 484
  Male | 859 | 858 | 1717
Race/Ethnicity, Customized [Number; unit: participants]
  White | 888 | 875 | 1763
  Black or African American | 33 | 36 | 69
  Hispanic | 141 | 136 | 277
  Other | 39 | 53 | 92
Current cigarette smoker [Number; unit: participants]
  Current Cigaratte Smoker | 428 | 431 | 859
  Non-Smoker | 664 | 660 | 1324
  Unknown | 9 | 9 | 18
Prior History of Characteristics and Risk Factors [Number; unit: participants] — Some study participants had more than one characteristic/risk factor and may be counted more than once.
  participants
    Angina | 240 | 255 | 495
    Myocardial infarction | 129 | 118 | 247
    Cerebrovascular disease | 48 | 34 | 82
    Peripheral-vessel disease | 44 | 39 | 83
    Heart Failure | 27 | 25 | 52
    PCI | 51 | 54 | 105
    CABG | 5 | 4 | 9
    Diabetes | 203 | 251 | 454
    Diabetes - Insulin Use | 63 | 61 | 124
    Hypertension | 528 | 543 | 1071
Infarct-related artery [Number; unit: participants] — Angiographic characteristic
  participants
    Left anterior descending coronary artery | 383 | 410 | 793
    Left circumflex coronary artery | 177 | 158 | 335
    Right coronary artery | 541 | 532 | 1073
Interval between MI and randomization [Median (Inter-Quartile Range); unit: days] | 8 [5 to 16] | 8 [5 to 17] | 8 [5 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Had a First Occurrence of the Primary End Point (Composite of Death From Any Cause, Nonfatal MI, or Class IV HF)
Description: Number of Patients with Events (death from any cause, nonfatal reinfarction, and hospitalization for New York Heart Association (NYHA) Class IV congestive heart failure). Events were centrally adjudicated.
Time Frame: Measured over a maximum 9-year follow-up period - 6 year median
Measure: Number; unit: participants
Arm/Group | Percutaneous Coronary Intervention Group | Medical Therapy Group
Number analyzed (Participants) | 1101 | 1100
participants | 230 | 219

2. Secondary Outcome: Number of Participants With Secondary Outcomes (Safety Events)
Description: Number of Participants with Secondary Outcomes (death from any cause, nonfatal MI, class IV HF, cardiac death, occurrence of selected clinical outcomes including stroke, hospitalization for CHF, sustained ventricular tachycardia/ventricular fibrillation, ICD implantation, or the composite end point). Events were centrally adjudicated.
Time Frame: Measured over a maximum 9-year follow-up period - 6 year median
Measure: Number; unit: participants
Arm/Group | Percutaneous Coronary Intervention Group | Medical Therapy Group
Number analyzed (Participants) | 1101 | 1100
participants
  Death from all causes | 150 | 153
  Fatal and nonfatal reinfarction | 77 | 65
  Nonfatal reinfarction | 75 | 61
  NYHA class IV heart failure (HF) | 51 | 53
  Cardiovascular death | 77 | 81
  Death or nonfatal reinfarction | 212 | 199
  NYHA class III or IV HF | 76 | 74
  Death, reinfarction, or NYHA class III or IV HF | 249 | 235
  Stroke | 29 | 24

ADVERSE EVENTS:
Arm/Group | Percutaneous Coronary Intervention Group | Medical Therapy Group
Serious Adverse Events (participants affected / at risk) | 226/1101 | 227/1100
Other Adverse Events (participants affected / at risk) | 75/1101 | 61/1100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention Group (N=1101) | Medical Therapy Group (N=1100)
Death from all causes (Cardiac disorders) | 150 (150) | 153 (153)
NYHA class III or IV Heart Failure (Cardiac disorders) | 76 (76) | 74 (74)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention Group (N=1101) | Medical Therapy Group (N=1100)
Nonfatal reinfarction (Cardiac disorders) | 75 (75) | 61 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The NIH Public Access Policy ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication. To help advance science and improve human health, the Policy requires that these papers are accessible to the public on PubMed Central no later than 12 months after publication.